CLINICAL TRIAL: NCT02906059
Title: A Phase Ib Study Combining Irinotecan With AZD1775, a Selective Wee 1 Inhibitor, in RAS (KRAS or NRAS) or BRAF Mutated Metastatic Colorectal Cancer Patients Who Have Progressed on First Line Therapy
Brief Title: Study of Irinotecan and AZD1775, a Selective Wee 1 Inhibitor, in RAS or BRAF Mutated, Second-line Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-01168
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: RAS; KRAS; NRAS; BRAF; Mutated; Wee1 inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — adavosertib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD1775 & Irinotecan (Experimental): Group AZD1775 (study drug); Irinotecan (chemotherapy)
  1) 125 mg two times a day (BID) for 3 days every 2 weeks; 180mg/m2 every 2 weeks
  2A) 150 mg BID for 3 days every 2 weeks; 180mg/m2 every 2 weeks
  2B) 125 mg BID for 5 days every 2 weeks; 180mg/m2 every 2 weeks
  3) 150 mg BID for 5 days every 2 weeks ; 180mg/m2 every 2 weeks
  Interventions: Drug: AZD1775; Drug: Irinotecan

INTERVENTIONS:
Drug: AZD1775
Drug: Irinotecan
  Other Names: Camptosar, Campto

SUMMARY:
The purpose of this study is to determine whether combination therapy of irinotecan with AZD1775 is safe and effective in treating mutated metastatic colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent prior to any study specific procedures
* Age 18 years or older
* Histological or cytological confirmation of Colorectal Cancer (CRC) with available tissue, currently stage IV
* Failure of first-line anti-cancer therapy with an oxaliplatin and bevacizumab based regimen (either radiological documentation of disease progression or due to toxicity) or subsequent relapse of disease following first-line therapy. Patients relapsing within 12 months of completing adjuvant FOLFOX will also be considered eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 1
* At least one lesion, not previously irradiated, that can be accurately measured as ≥ 10 mm in the longest diameter (LD) with spiral computed tomography (CT) scan or as ≥ 20 mm with conventional techniques (conventional CT, MRI) and which is suitable for accurate repeated measurements
* Tumor sample confirmed as KRAS or NRAS [codons 12 and 13 (exon 2), 59 and 61 (exon 3), and 117 and 146 (exon 4)] or BRAF [codon 600 (exon 15)] mutation positive.
* Patients must be able to swallow AZD1775 capsules

Exclusion Criteria:

* Treatment within 14 days prior to first study treatment with conventional therapy or treatment within 28 days prior to first study treatment with an investigational drug
* Received more than 1 line of systemic treatment for advanced/metastatic CRC and/or a patient whose first line therapy did not contain oxaliplatin and bevacizumab
* Prior treatment with a Wee1 inhibitor or any irinotecan containing regimen
* Any unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy, except for alopecia and neurotoxicity.
* The last radiation therapy within 4 weeks prior to starting study treatment, or limited field of radiation for palliation within 2 weeks of the first dose of study treatment
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) which would prevent administration of study treatment
* History of hypersensitivity to AZD1775, irinotecan, or any excipients of these agents
* Brain metastases or spinal cord compression unless asymptomatic, treated and stable off steroids and anti-convulsants for at least 3 months
* Laboratory values as listed below (from laboratory results during screening):

  * Absolute Neutrophil Count (ANC) <1.5 x 10^9/L (1500 per mm3)
  * Platelets < 100 x 109/L (100,000 per mm3)
  * Hemoglobin <9.0 g/dL
  * Serum bilirubin >Upper Limit of Normal (ULN)
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT):

    * > 2.5 x ULN
    * > 5 x ULN, if liver metastasis present
  * Creatinine clearance < 50 cc/min measured or calculated by Cockcroft Gault equation - Cardiac conditions as follows:
  * Uncontrolled hypertension (BP ≥ 170/100 despite optimal therapy)
  * Heart failure New York Heart Association (NYHA) Class II or above
  * Prior or current cardiomyopathy
  * If NYHA Class I heart failure, Left Ventricular Ejection Fraction (LVEF) by Multi Gated Acquisition Scan (MUGA) or Echocardiogram (ECHO) is less than 50%
  * Unstable ischemic heart disease (myocardial infarction within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly)
  * Mean resting corrected QT (QTc) interval using the Fridericia formula (QTcF) > 450 msec/male and > 470 msec/female (as calculated per institutional standards) obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart at study entry, or congenital long QT syndrome
  * Patients with significant ventricular or supraventricular arrhythmias and patients with cardiac conduction abnormalities that are not controlled (e.g. with a pacemaker or medication).
* Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate ingestion and absorption of an oral agent
* Clinical evidence of bowel obstruction at the time of study entry
* Female patients who are pregnant or breast-feeding, or male or female patients of reproductive potential who are not employing an effective method of birth control
* History of another primary malignancy within 5 years prior to starting study treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ. Patients with an early stage cancer, now off therapy for at least 3 years may be enrolled with permission of the PI if that disease is unlikely to interfere with the primary endpoints of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09; Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Number of participants dose limiting toxicities with treatment-related adverse events as assessed by common terminology criteria for adverse events (CTCAE), version 4. | Up to 12 months

SECONDARY OUTCOMES:
Tumor assessment by imaging techniques using Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 | From baseline to every 8 weeks up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Cohen, MD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- Laura and Isaac Perlmutter Cancer Center, New York, New York, United States